CLINICAL TRIAL: NCT02406820
Title: Characterizing Noninvasive Cardiovascular Measures Collected Passively and In Response to an Isometric Handgrip Stress Test From CVInsight®, Connex ProBP, and Zio® XT Patch in Patients With Acute Decompensated Heart Failure
Brief Title: Correlating Noninvasive Cardiovascular Measures to Left Ventricular End Diastolic Pressure in Heart Failure
Status: Terminated | Type: Observational
Why Stopped: Strategic closure by sponsor to pursue other indications.
Sponsor: Intelomed, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: HF001
Record Dates: First submitted 2015-03-26; First posted 2015-04-02 (Estimated); Last update posted 2016-08-30 (Estimated); Status verified 2016-08

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- No Indwelling PAC, Daily Testing: Acutely decompensated heart failure patients undergoing a right heart catheterization for whom a retained indwelling PAC is not clinically indicated and who are registered to twice daily non-invasive hemodynamic monitoring during an isometric handgrip stress test (IHGST).
  Interventions: Device: Non-invasive hemodynamic monitoring (CVInsight™ [CVI])
- Indwelling PAC, Daily Testing: Acutely decompensated heart failure patients undergoing a right heart catheterization for whom a retained indwelling PAC is clinically indicated and who are registered to three times daily non-invasive hemodynamic monitoring during an isometric handgrip stress test (IHGST).
  Interventions: Device: Non-invasive hemodynamic monitoring (CVInsight™ [CVI])
- No Indwelling PAC, No Daily Testing: Acutely decompensated heart failure patients undergoing a right heart catheterization for whom a retained indwelling PAC is clinically indicated and who are registered to no daily non-invasive hemodynamic monitoring during an isometric handgrip stress test (IHGST).
  Interventions: Device: Non-invasive hemodynamic monitoring (CVInsight™ [CVI])

INTERVENTIONS:
Device: Non-invasive hemodynamic monitoring (CVInsight™ [CVI])

SUMMARY:
HF001 is a prospective observational study utilizing non-invasive medical devices that may be able to discriminate changes in heart failure while acutely decompensated patients undergo routine interventional therapies in a hospital setting. Subjects will be monitored using CVInsight™ [CVI] via a finger and/or forehead sensor, while performing an isometric handgrip stress test (IHGST). Changes in the CVI signal will be analyzed and correlated to standard assessments of heart failure including pulmonary artery catheter (PAC) pressures, blood pressure (BP), patient symptoms, and physical exam findings. The results of this study will be used to develop a powered study to determine if a new configuration of non-invasive monitoring devices can be used to monitor heart failure status more sensitively than current non-invasive techniques.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ≥ 18 years old
* Signs and symptoms of congestive heart failure including two of the following:
* Peripheral edema (e.g. abdominal distension, hepatomegaly, lower extremity edema) in the setting of elevated jugular venous pressure as assessed by the clinical examination, or by right heart catheterization.
* Pulmonary edema or pleural effusion as seen on chest X-ray
* Elevated N-terminal pro-brain natriuretic peptide (NT-Pro BNP) 2x the upper limit of normal.
* Willing and able to comply with the study protocol
* Willing and able to give valid Informed Consent

Exclusion Criteria:

* Pregnant patients
* Presence of Left Ventricular Assist Device (LVAD) or heart transplant
* Complex congenital heart disorder or prosthetic valve on right side
* Known mitral stenosis
* Unstable medical condition or impairment other than condition associated with HF
* Unstable hypertension
* Too unstable in the judgment of the investigator to be included in the study
* Active lung infection or acute pulmonary decompensation
* Elevated white blood cell count and signs of infection are evident
* Does not have the cognitive ability to understand and sign the Informed Consent
* Does not have the cognitive capacity to perform handgrip test
* Is not able to perform a handgrip stress test
* Is not able to wear any of the devices
* Patient's life expectancy is less than 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acutely decompensated heart failure patients admitted to acute care setting, who require a right heart catheterization.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2015-04; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Evidence of correlation between CVInsight signals and Pulmonary Capillary Wedge Pressure or Pulmonary Artery Pressure | Upon completion of catheter assessments for all enrolled subjects, approximately 6 months from study activation

CONTACTS AND LOCATIONS:
Overall Officials: David Majure, MD, Principal Investigator — MedStar Health
Locations (1):
- Medstar Washington Hospital Center, Washington D.C., District of Columbia, United States